CLINICAL TRIAL: NCT00529971
Title: A Randomized Controlled Trial of a Mindfulness-Based Stress Reduction Intervention for Men Living With HIV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other); Canadian Foundation for AIDS Research (CANFAR) (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 015005
Record Dates: First submitted 2007-09-11; First posted 2007-09-14 (Estimated); Last update posted 2007-10-03 (Estimated); Status verified 2007-09

CONDITIONS: HIV Infections
Keywords: Mindfulness; HIV; Male; Living with HIV; 18-70 years of age; live within one hour of hospital; fluent in English; Complementary Therapies; HIV Therapeutic Vaccine
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Participants in the first arm participate in an 8-week MBSR group
  Interventions: Behavioral: MBSR group
- 2 (Active Comparator): Participants assigned to the control arm do not receive the MBSR program but may or may not be receiving current psychotherapy or counselling
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: MBSR group — 8-week MBSR group, 3 hours per week plus one all day retreat
  Arms: 1
Other: Control — Treatment as usual, which could include medications or psychotherapy
  Arms: 2

SUMMARY:
This study will examine the effectiveness of Mindfulness-Based Stress Reduction (MBSR) in helping men living with HIV cope with negative emotions and stresses in their life. MBSR is an approach to reducing stress for patients with chronic medical conditions. It involves systematic training in mindfulness meditation practices to increase quality of life and to reduce general stress, anxiety, depression or pain. The effectiveness of MBSR will be evaluated by looking at changes in participants' experience of stress, anxiety associated with pain management and psychosocial functioning before and after they receive the MBSR compared with participants who do not receive the MBSR treatment.

In order to participate, individuals must be: male, living with HIV, age 18-70 years, live within one hour of participating centre, and have a good understanding of the English language. Questionnaires will be completed before individuals begin the program, at the end of the intensive phase (8 weeks) and at 6 months after the start of the group program. The primary program evaluation outcome will be a reduction in stress; secondary evaluation outcomes will include the improvements in the physical and emotional experience of pain as well as general psychosocial functioning and self-esteem.

DETAILED DESCRIPTION:
In most health care settings, psychosocial interventions that target stress and distress states that are integrated into routine HIV care will need to serve a large number of patients. Due to their time- and cost- efficiency, group approaches are being used increasingly in medical settings to address this need. One approach that has been used successfully in cancer and other chronic diseases is mindfulness-based stress reduction (MBSR), an 8-week manualized treatment program that provides mood management techniques based on training in mindfulness, a metacognitive skill. A recent randomized controlled trial in cancer demonstrated that this brief intervention significantly reduced anxiety and depression symptoms and that these gains were maintained at a six-month follow-up. Similar results have been obtained in a heterogeneous sample of medical patients. Although research in this area is in its infancy, it does appear that MBSR may be effective in the management of anxiety and mood symptoms that are common across various medical conditions and thus may be a good treatment option in men living with HIV.

Preliminary evidence, gathered from a pilot assessment of an MBSR program for HIV positive men, demonstrated significant pre- to post-intervention reductions in anxiety and depression, as well as overall mood disturbance scores on standardized measures, and thus, MBSR has promise in this population. A randomized controlled trial is clearly needed however before can be recommended as a psychosocial treatment for men with HIV. It is predicted that MBSR will be effective in mitigating anxiety and depressive symptoms, as well as HIV-related distress, among HIV patients (Hypothesis #1).

MBSR appears to be particularly well suited for anxiety- and depression- spectrum symptoms because it targets cognitive processes that contribute to and maintains them. Current cognitive models emphasize the central role of worry and rumination in the onset and maintenance of anxiety and depression, respectively. Worry can perpetuate an upward spiral of increased emotional arousal and intrusive thoughts heightening anxiety symptoms. Similarly, rumination can escalate a spiraling cycle of dysphoric affect and associated negative thinking that can lead eventually to a major depressive episode. (MBSR utilizes training in attention regulation that is thought to provide patients with a skill that enables them to disengage from patterns of worry and rumination that otherwise would perpetuate negative affect. Consistent with this prediction, Dr. Bishop (co-investigator) has found evidence from a recently completed pilot study that mindfulness training results in decreased frequency of worry and rumination. Although preliminary, MBSR may be associated with decreases in both worry and rumination (Hypothesis #2) and that, consistent with current cognitive models, decreases in worry and rumination would moderate the reductions in anxiety and depression, respectively (Hypothesis #3).

We are also interested in whether this approach is effective for the management of pain, which is prevalent in this population. There is substantial evidence that anxiety, and particularly pain-related fear, can heighten the perception of the intensity and unpleasantness of pain and that anxiety management can lessen pain. Since we anticipate that MBSR will reduce anxiety in this study, we would further expect that it would also reduce the subjective experience of pain (Hypothesis #4). There is some evidence from an uncontrolled trial suggesting that MBSR may be highly effective for managing chronic pain. If MBSR can be used to effectively mitigate pain, then this too would have a recursive effect on mood. Pain in medical populations is a significant factor in emotional distress and psychiatric morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Living with HIV
* 18-70 years of age
* Fluent in English
* Lives within one hour of the hospital

Exclusion Criteria:

* Severe depression
* Current suicide ideation
* Substance abuse
* Impaired cognitive function

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2003-12; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Subjects in the MBSR group will have greater improvement in measures of psychosocial functioning (i.e. anxiety, depression, HIV-related distress, affectivity) at 8 weeks and 6-months post-intervention | 8 weeks and 6 months after start of intervention
Subjects in the MBSR group will demonstrate significantly greater improvement on measures of worry and rumination at 8 weeks and 6-months post-intervention | 8 weeks and 6 months after start of intervention
MBSR will result in greater improvement in pain compared to the control arm | 8 weeks and 6 months after start of intervention

SECONDARY OUTCOMES:
Reductions in anxiety and depression during MBSR will be moderated by reductions in worry and ruminations, respectively | 8 weeks and 6 months after start of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Bill Gayner, M.S.W., Principal Investigator — MOUNT SINAI HOSPITAL; Mary Jane Esplen, Ph.D., Principal Investigator — University Health Network, Toronto
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada